CLINICAL TRIAL: NCT04914741
Title: A Multicentre Trial of Frontline R-CHOP/Pola-RCHP and Glofitamab in Younger, Higher Risk Patients With Diffuse Large B Cell Lymphoma (DLBCL)
Brief Title: A Multicentre, Parallel Arm, Open-label Trial of Frontline R-CHOP/Pola-RCHP and Glofitamab in Younger, Higher Risk Patients With Diffuse Large B Cell Lymphoma (DLBCL)
Acronym: COALITION
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/047
Record Dates: First submitted 2021-05-24; First posted 2021-06-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma
Keywords: DLBCL; HGBL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisolone; glofitamab; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glofitamab plus R-CHOP (Experimental): Participants will receive treatment in 21 day cycles consisting of R-CHOP in cycle 1, followed by R-CHOP plus glofitamab for cycles 2-6, and two cycles of glofitamab monotherapy consolidation. Patients may also receive high-dose methotrexate CNS prophylaxis at investigator discretion.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisolone; Drug: Glofitamab
- Glofitamab plus polatuzumab vedotin-RCHP (Experimental): Participants will receive treatment in 21 day cycles consisting of R-CHOP in cycle 1, followed by polatuzumab vedotin-RCHP plus glofitamab for cycles 2-6, and two cycles of glofitamab monotherapy consolidation. Patients may also receive high-dose methotrexate CNS prophylaxis at investigator discretion.
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisolone; Drug: Glofitamab; Drug: Polatuzumab vedotin

INTERVENTIONS:
Drug: Rituximab — Rituximab 375 mg/m^2 administered by IV infusion on Day 1 of every 21-day cycle
Drug: Cyclophosphamide — Cyclophosphamide 750mg/m^2 administered by IV infusion on Day 1 of every 21-day cycle
Drug: Doxorubicin — Doxorubicin 50mg/m^2 administered by IV infusion on Day 1 of every 21-day cycle
Drug: Vincristine — Vincristine 1.4mg/m^2 administered by IV infusion on Day 1 of every 21-day cycle
  Arms: Glofitamab plus R-CHOP
Drug: Prednisolone — Prednisolone 100mg orally on Days 1-5 of every 21-day cycle
Drug: Glofitamab — Glofitamab will be administered by IV infusion as per the schedule specified in the respective arm
  Other Names: RO7082859; CD20-TCB
Drug: Polatuzumab vedotin — Polatuzumab 1.8mg/kg administered by IV infusion on Day 1 of every 21-day cycle
  Arms: Glofitamab plus polatuzumab vedotin-RCHP

SUMMARY:
This is an open label, multi-centre, phase Ib/II, parallel arm study evaluating the safety and tolerability of glofitamab in addition to backbone chemotherapy consisting of R-CHOP or polatuzumab vedotin-RCHP for younger patients with higher-risk Diffuse Large B-cell Lymphoma or High Grade B-Cell Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18yo and ≤65yo at the time of signing consent
2. Have a histologically confirmed diagnosis of one of the following, according to the 2016 WHO classification:

   1. DLBCL, NOS or DLBCL arising as a result of transformation of an indolent lymphoma
   2. HGBL, NOS
   3. HGBL with rearrangements of MYC and BCL2 and/or BCL6
3. For DLBCL, and HGBL, NOS meets one of the following risk criteria:

   a. NCCN-IPI of ≥4 or IPI ≥3 (appendix 1 and 3)
4. Considered fit for 6 cycles of full dose R-CHOP chemotherapy, as per the Investigator
5. ECOG performance status (appendix 5) of:

   1. 0-2 inclusive or 3 if directly attributable to lymphoma for patients entering the trial prior to cycle 1 of R-CHOP
   2. 0-1 inclusive for patients entering the trial at cycle 2
6. Patients must be treatment-naïve or have received a maximum of one cycle of full-dose R-CHOP chemotherapy (with or without a steroid pre-phase)
7. Able to provide an archival pre-treatment biopsy.
8. Have measurable disease on a pre-chemotherapy PET/CT, defined as at least one bi-dimensionally measurable nodal lesion of >1.5cm in longest dimension, or at least one bi-dimensionally measurable extranodal lesion of >1.0cm in longest dimension
9. Life expectancy (in the opinion of the Investigator) of ≥ 18 weeks
10. Adequate haematological function
11. Adequate renal function
12. Adequate hepatic function
13. Negative serologic or PCR test results for active acute or chronic HBV infection.
14. Non-haematological AEs from prior anti-cancer therapy must have resolved to Grade ≤1 (with the exception of alopecia and inclusion criteria 10-12)
15. Negative test results for HCV and HIV.

Exclusion Criteria:

1. Inability to comply with protocol mandated hospitalisations and restrictions
2. Prior systemic treatment of an underlying indolent lymphoma with an anthracycline-containing regimen
3. Richter's syndrome
4. Patients with known CNS involvement by lymphoma
5. With the exception of rituximab, any prior treatment with systemic immunotherapeutic agents, including, but not limited to, radio-immuno-conjugates, antibody-drug conjugates, immune/cytokines, and monoclonal antibodies within 4 weeks or five half-lives of the drug, whichever is shorter, before the first dose of study drug
6. With the exception of CHOP used as a first cycle of lymphoma treatment, any chemotherapeutic agent, or treatment with any other investigational agent within 4 weeks prior to study treatment
7. Prior solid organ transplantation
8. Prior autologous or allogeneic stem cell transplantation
9. A history of treatment-emergent immune related AEs associated with prior immunotherapeutic agents
10. Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease

    1. Note: patients with a history of stroke who have not experienced a stroke or transient ischaemic attack in the past 2 years are allowed
    2. Note: patients with a history of epilepsy who have not experienced a seizure in the past 2 years are allowed, so long as continuation of any ongoing established pharmacologic treatment is not contraindicated
11. Past history of confirmed progressive multifocal leukoencephalopathy
12. Past history of chronic active EBV or HLH
13. Major surgery or significant traumatic injury <28 days prior to study treatment or anticipation of the need for major surgery during study treatment
14. Significant cardiovascular disease, defined as:

    1. A left ventricular ejection fraction (as determined by nuclear gated blood pool scan or echocardiogram) <50%
    2. Myocardial infarction or unstable angina within the past 6 months
    3. Unstable arrhythmia
    4. Any other cardiac illness that, in the opinion of the Investigator or CPI, makes the patient unsuitable for anthracycline containing therapy
15. Significant pulmonary disease, including but not limited to clinically significant obstructive pulmonary disease or history of bronchospasm
16. Current grade >1 peripheral neuropathy by clinical examination or demyelinating form of Charcot-Marie-Tooth disease
17. Known clinically significant liver disease, including active viral or other hepatitis, current alcohol abuse, or cirrhosis
18. Administration of a live, attenuated vaccine within 4 weeks before study treatment note: influenza vaccination should be given during influenza season only. Patients must not receive live, attenuated influenza vaccine at any time during the study treatment period
19. History of other active malignancy within 5 years prior to registration, with the exception of:

    1. FL or MZL, previously untreated, or treated with no more than one line of therapy which must not have contained an anthracycline
    2. Basal or squamous cell carcinoma or Stage 1 melanoma of the skin or in situ carcinoma of the cervix
    3. Prior malignancy treated with a curative intent that has remained in remission without treatment for ≥2 years prior to registration
20. Patients with known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of the nail beds) at registration

    a. Note: Patients with latent tuberculosis are excluded
21. Other significant life-threatening illness or medical condition which, in the Investigator's opinion, could compromise the patient's safety, interfere with absorption or metabolism of study drug, affect compliance with the protocol or interpretation of results, or put the study outcomes at undue risk
22. Major contraindication to any of the individual components of the chemotherapy backbone (R, C, H, O, Polatuzumab vedotin, prednisolone)
23. Patients who are pregnant or breastfeeding

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
To assess safety of the combination of glofitamab and R-CHOP or pola-RCHP according to number of participants with treatment-related adverse events | From start of treatment till the end of study, assessed up to approximately 60 months
To evaluate the Relative Dose Intensity (RDI) of the chemotherapy backbone | From start of study treatment till the end of study treatment, assessed up to approximately 12 months
To evaluate the rates of early chemotherapy discontinuation | From start of study treatment till the end of study treatment, assessed up to approximately 12 months

SECONDARY OUTCOMES:
To estimate the proportion of patients achieving a complete response (CR) after cycles 2, 4 and at end of induction treatment (6 cycles) of the novel combination therapy according to Lugano 2014 criteria | Up to approximately 6 months (each cycle is 21 days)
To estimate overall response rate (ORR) | Up to approximately 6 months (each cycle is 21 days)
To describe progression free survival (PFS) | From first dose of chemotherapy induction to first date of objectively documented progressive disease or date of death of any cause, whichever occurs first, assessed up to approximately 60 months
To describe the duration of response (DoR) measured in the subset of patients who achieved CR or PR | Time from the first documented disease response to the date of progressive disease or death, whichever occurs first, assessed up to approximately 60 months
Overall survival (OS) as defined as the time from first dose of chemotherapy induction to the date of death from any cause | From first dose of chemotherapy induction to the date of death from any cause, assessed up to approximately 60 months

OTHER OUTCOMES:
Correlation between circulating tumour DNA detection and response (CR and ORR) | From start of treatment till end of study assessed up to 60 months
Comparison of efficacy (rates of CR, ORR, DOR, PFS and OS) between the two study arms | From start of treatment till end of study assessed up to 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Principal Investigator — Peter MacCallum Cancer Centre & Royal Melbourne Hospital
Locations (15):
- Australia (15):
  - Concord Repatriation General Hospital, Camperdown, New South Wales
  - St Vincent's Public Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Princess Alexander Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Barwon Health, Geelong, Victoria
  - Cabrini Hospital, Malvern, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St Vincent's Hospital Melbourne, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Epworth Healthcare, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Minson A, Verner E, Giri P, Butler J, Janowski W, Cheah CY, Ratnasingam S, Wong SM, Ku M, Hertzberg M, Herbert K, Hamad N, Yannakou CK, Swain F, Neeson P, Steiner TM, Saghebi J, Blombery P, Hunter SM, Robertson M, Lau LS, Bennett R, Harrop S, Xie J, Seymour JF, Dickinson MJ. Glofitamab Combined With Pola-R-CHP or R-CHOP as First Therapy in Younger Patients With High-Risk Large B-Cell Lymphoma: Results From the COALITION Study. J Clin Oncol. 2025 Aug 10;43(23):2595-2605. doi: 10.1200/JCO-25-00481. Epub 2025 Jun 18. PMID 40532125